CLINICAL TRIAL: NCT04209777
Title: Clinical Evaluation of Smoker Periodontal Subjects After Lactobacillus-reuteri Probiotics and Antibiotics Therapy With Scaling and Root Debridement: a Clinical Trial
Brief Title: Clinical Evaluation of Smoker Periodontal Subjects After Lactobacillus-reuteri Probiotics and Antibiotics Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mehwish Ghazal, Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGhazal
Record Dates: First submitted 2019-12-18; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Periodontal Diseases; Smoking
MeSH Terms: conditions — Periodontal Diseases; Smoking | interventions — Tooth Exfoliation; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotics (Active Comparator): The antibiotic group is provided with amoxicillin capsules 500mg and metronidazole tablets 400mg three times a day for 7 days along with the placebo of probiotics twice daily for 30 days.
  Interventions: Drug: Antibiotics
- Probiotics (Experimental): The probiotic group is provided with Lactobacillus-reuteri probiotics (2x10(8)CFU) twice daily after brushing for 30 days.
  Interventions: Drug: Probiotic Blend Chewable Tablet

INTERVENTIONS:
Drug: Probiotic Blend Chewable Tablet — Lactobacillus-reuteri probiotics were used as an experimental drug.
  Other Names: Scaling and root debridement.
  Arms: Probiotics
Drug: Antibiotics — Amoxicillin capsules 500mg and metronidazole tablets 400mg antibiotics were used as an active comparator.
  Other Names: Scaling and root debridement.
  Arms: Antibiotics

SUMMARY:
It is a clinical trial conducted on smokers with chronic periodontitis in which the participants are divided into two groups and one group is provided with antibiotics while the other with probiotics as an adjunct to non-surgical therapy. The participants were assessed for change in probing pocket depths, attachment loss, bleeding on probing, plaque index and gingival index after 1-month and 3-month period.

DETAILED DESCRIPTION:
Background:

Periodontal disease is a chronic inflammatory disease of the supporting structures of the tooth which includes periodontal ligament, cementum, and bone. Conventional periodontal therapy involves a non-surgical and surgical method for mechanical debridement of supragingival and subgingival sites to eliminate the pathogens and reduce inflammation of the periodontium. Smokers respond less to conventional therapy and require antibiotics for additional benefits. Where the use of antibiotics provides benefits to the host, the increasing proportion of developing antibiotic resistance are a major concern. The introduction of "Probiotics" as a treatment option is under special consideration. According to WHO, Probiotics are defined as viable micro-organisms which when delivered in an appropriate dose, provides health benefits. Lactobacillus-reuteri has been considered as a reliable option in regards to safety with no reported adverse effects, in the treatment of periodontitis as an adjunct to Scaling and Root Debridement.

Objectives:

The objective of the present study is to evaluate the clinical improvement of Lactobacillusreuteri Probiotics in comparison to a combination of amoxicillin and metronidazole antibiotics in smokers with moderate to severe chronic periodontitis after non-surgical scaling and root debridement.

Method:

A total number of 60 Smokers with moderate to severe chronic periodontitis were randomized into two groups after taking consent. Group 1 received amoxicillin and metronidazole for 7 days and placebo for Probiotics for 30 days. Group 2 was provided with 1 tablet of Lactobacillus-reuteri Probiotics (2x108CFU) twice daily after brushing for 30 days and a placebo for antibiotics for 7 days. At recruitment, scaling and root debridement were performed and change in pocket depth, attachment loss, gingival index, plaque index and bleeding on probing were recorded. The same outcomes were recorded again at 1 month and 3 months follow-up. Mean, standard deviation and confidence interval were reported using SPSS version-20.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy males or females.
* at least 35 years of age with minimal 3 natural teeth in each quadrant excluding 3rd molar.
* previously untreated moderate to severe generalized chronic periodontitis
* were current smokers having ≥10 cigarettes /day.

Exclusion Criteria:

* having periodontal therapy within the past 6 months.
* have undergone antibiotics or long-term NSAIDS therapy within the past 6 months.
* have an allergy to penicillin and metronidazole.
* having either fixed or removable prosthesis.
* pregnant or nursing females.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-07-08 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Change in Probing pocket depth | At baseline.
  Probing pocket depth is recorded on six sites per tooth.
Change in Probing pocket depth | After 1-month.
  Probing pocket depth is recorded on six sites per tooth.
Change in Probing pocket depth | After 3-months.
  Probing pocket depth is recorded on six sites per tooth.
Change in Clinical attachment level | At baseline.
  Clinical attachment level is recorded on six sites per tooth.
Change in Clinical attachment level | After 1-month.
  Clinical attachment level is recorded on six sites per tooth.
Change in Clinical attachment level | After 3-months.
  Clinical attachment level is recorded on six sites per tooth.
Change in Bleeding on probing | At baseline.
  Bleeding on probing is recorded on six sites per tooth. Presence or absence of bleeding is checked.
Change in Bleeding on probing | After 1-month.
  Bleeding on probing is recorded on six sites per tooth. Presence or absence of bleeding is checked.
Change in Bleeding on probing | After 3-months.
  Bleeding on probing is recorded on six sites per tooth. Presence or absence of bleeding is checked.

SECONDARY OUTCOMES:
Change in Plaque index | At baseline.
  Plaque index is recorded to check deposits on six teeth which are left upper first molar, upper left lateral incisor, upper right premolar, and lower right first molar, lower right lateral incisor and lower left premolar. all the six sites of each tooth are examined.
  0= No plaque; 1= A film of plaque adhering to the free gingival margin and adjacent area of the tooth; 2= Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye; 3= Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Change in Plaque index | After 1-month.
  Plaque index is recorded to check deposits on six teeth which are left upper first molar, upper left lateral incisor, upper right premolar, and lower right first molar, lower right lateral incisor and lower left premolar. all the six sites of each tooth are examined.
  0= No plaque; 1= A film of plaque adhering to the free gingival margin and adjacent area of the tooth; 2= Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye; 3= Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Change in Plaque index | After 3-months.
  Plaque index is recorded to check deposits on six teeth which are left upper first molar, upper left lateral incisor, upper right premolar, and lower right first molar, lower right lateral incisor and lower left premolar. all the six sites of each tooth are examined.
  0= No plaque; 1= A film of plaque adhering to the free gingival margin and adjacent area of the tooth; 2= Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye; 3= Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Change in Gingival index | At baseline.
  Gingival index is recorded on six teeth which are left upper first molar, upper left lateral incisor, upper right premolar, and lower right first molar, lower right lateral incisor and lower left premolar. mesio-buccal, disto-buccal, buccal/facial margin and lingual gingival margin is assessed.
  0= Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
Change in Gingival index | After 1-month.
  Gingival index is recorded on six teeth which are left upper first molar, upper left lateral incisor, upper right premolar, and lower right first molar, lower right lateral incisor and lower left premolar. mesio-buccal, disto-buccal, buccal/facial margin and lingual gingival margin is assessed.
  0= Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
Change in Gingival index | After 3-months.
  Gingival index is recorded on six teeth which are left upper first molar, upper left lateral incisor, upper right premolar, and lower right first molar, lower right lateral incisor and lower left premolar. mesio-buccal, disto-buccal, buccal/facial margin and lingual gingival margin is assessed.
  0= Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Shahbaz Ahmed, BDS/FCPS, Study Director — Dow University of Health Sciences
Locations (1):
- Mehwish Ghazal, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The data will be available for sharing after 6-months of publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after the publication of the study for 1 year.
Access Criteria: Contact the principal investigator through email.

REFERENCES:
- [Result] Ikram S, Hassan N, Baig S, Borges KJJ, Raffat MA, Akram Z. Effect of local probiotic (Lactobacillus reuteri) vs systemic antibiotic therapy as an adjunct to non-surgical periodontal treatment in chronic periodontitis. J Investig Clin Dent. 2019 May;10(2):e12393. doi: 10.1111/jicd.12393. Epub 2019 Jan 20. PMID 30663271
- [Result] Morales A, Carvajal P, Silva N, Hernandez M, Godoy C, Rodriguez G, Cabello R, Garcia-Sesnich J, Hoare A, Diaz PI, Gamonal J. Clinical Effects of Lactobacillus rhamnosus in Non-Surgical Treatment of Chronic Periodontitis: A Randomized Placebo-Controlled Trial With 1-Year Follow-Up. J Periodontol. 2016 Aug;87(8):944-52. doi: 10.1902/jop.2016.150665. Epub 2016 Mar 4. PMID 26944407
- [Result] Theodoro LH, Claudio MM, Nuernberg MAA, Miessi DMJ, Batista JA, Duque C, Garcia VG. Effects of Lactobacillus reuteri as an adjunct to the treatment of periodontitis in smokers: randomised clinical trial. Benef Microbes. 2019 Apr 19;10(4):375-384. doi: 10.3920/BM2018.0150. Epub 2019 Apr 1. PMID 30931588
- [Result] Vicario M, Santos A, Violant D, Nart J, Giner L. Clinical changes in periodontal subjects with the probiotic Lactobacillus reuteri Prodentis: a preliminary randomized clinical trial. Acta Odontol Scand. 2013 May-Jul;71(3-4):813-9. doi: 10.3109/00016357.2012.734404. Epub 2012 Nov 26. PMID 23176716
- [Result] Assem NZ, Alves MLF, Lopes AB, Gualberto EC Junior, Garcia VG, Theodoro LH. Antibiotic therapy as an adjunct to scaling and root planing in smokers: a systematic review and meta-analysis. Braz Oral Res. 2017 Jul 3;31:e67. doi: 10.1590/1807-3107BOR-2017.vol31.0067. PMID 28678975
- [Result] Grusovin MG, Bossini S, Calza S, Cappa V, Garzetti G, Scotti E, Gherlone EF, Mensi M. Clinical efficacy of Lactobacillus reuteri-containing lozenges in the supportive therapy of generalized periodontitis stage III and IV, grade C: 1-year results of a double-blind randomized placebo-controlled pilot study. Clin Oral Investig. 2020 Jun;24(6):2015-2024. doi: 10.1007/s00784-019-03065-x. Epub 2019 Oct 16. PMID 31620939
- [Result] Albandar JM. Adjunctive antibiotics with nonsurgical periodontal therapy improve the clinical outcome of chronic periodontitis in current smokers. J Evid Based Dent Pract. 2012 Sep;12(3 Suppl):63-6. doi: 10.1016/S1532-3382(12)70015-5. PMID 23253833
- [Result] Morales A, Gandolfo A, Bravo J, Carvajal P, Silva N, Godoy C, Garcia-Sesnich J, Hoare A, Diaz P, Gamonal J. Microbiological and clinical effects of probiotics and antibiotics on nonsurgical treatment of chronic periodontitis: a randomized placebo- controlled trial with 9-month follow-up. J Appl Oral Sci. 2018 Jan 18;26:e20170075. doi: 10.1590/1678-7757-2017-0075. PMID 29364340
- [Result] Ikram S, Hassan N, Raffat MA, Mirza S, Akram Z. Systematic review and meta-analysis of double-blind, placebo-controlled, randomized clinical trials using probiotics in chronic periodontitis. J Investig Clin Dent. 2018 Aug;9(3):e12338. doi: 10.1111/jicd.12338. Epub 2018 Mar 31. PMID 29604177